CLINICAL TRIAL: NCT03468387
Title: Primary Urethral Realignment vs. Suprapubic Cystostomy for Initial Management of Pelvic Fracture Urethral Injury in Children: Randomized Clinical Trial
Brief Title: Primary Urethral Realignment vs. Suprapubic Cystostomy for Initial Management of Pediatric Pelvic Fracture Urethral Injury
Acronym: PREvsSPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osama, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URSP
Record Dates: First submitted 2018-03-06; First posted 2018-03-16 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Urethral Injury
MeSH Terms: interventions — Cystostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary realignment (Active Comparator)
  Interventions: Procedure: Primary realignment
- Suprapubic cystostomy (Active Comparator)
  Interventions: Procedure: Suprapubic cystostomy

INTERVENTIONS:
Procedure: Primary realignment — Endoscopic realignment of rupture urethra over a urethral catheter
  Arms: Primary realignment
Procedure: Suprapubic cystostomy — Percutaneous cystostomy catheter will be inserted under sonographic guidance
  Arms: Suprapubic cystostomy

SUMMARY:
It is prospective randomized comparative clinical trial comparing primary urethral realignment vs. suprapubic cystostomy in initial management of pediatric pelvic fracture urethral injury regarding:

1. The success rate after initial intervention.
2. The need for urethroplasty in the failed realignment group and cystostomy group.
3. The success rate of urethroplasty in the failed realignment group and cystostomy group.

ELIGIBILITY:
Inclusion Criteria:

* Male children less than 18 years presenting with pelvic fracture urethral injury

Exclusion Criteria:

* Associated bladder neck injury.
* Associated rectal injury.
* Late presentation >2weeks since trauma.
* History of previous urethral intervention.

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
The success rate after initial intervention (realignment or suprapubic cystostomy). | 3 months after initial intervention.
  The fulfillment of success criteria after initial intervention which includes good stream, no postvoid residual urine, normal Qmax for age and free retrograde urethrogram

SECONDARY OUTCOMES:
The success rate of urethroplasty in both groups. | 3 months after urethroplasty.
  The surgical outcome of urethroplasty in cases of children with posterior urethral stricture after failed realignment or suprapubic cystostomy.
The need for urethroplasty in both groups. | 3 months after initial intervention
  Comparison of the need for urethroplasty in children with failed realignment or suprapubic cystostomy.